CLINICAL TRIAL: NCT06471348
Title: Postoperative Pain Control in AIS Using Liposomal Bupivacaine vs. 0.25% Bupivacaine
Brief Title: Postoperative Pain Control in AIS Using Liposomal Bupivacaine vs. 0.25% Bupivacaine With Epinephrine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Craig Birch, Instructor of Orthopedic Surgery, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-P00048597
Record Dates: First submitted 2024-05-21; First posted 2024-06-24 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Post Operative Pain; Spinal Fusion
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local infiltration with liposomal bupivacaine (Experimental): Patients randomized into the liposomal bupivacaine group will receive anesthesia and undergo standard posterior spinal fusion surgery. The local infiltration would occur in a single stage, after instrumentation and correction maneuver is performed, just prior to closure of the deep fascial layer. The dose would be injected via multiple small volume injections into the paraspinal musculature, spaced approximately 1 cm apart.
  Interventions: Drug: Bupivacaine liposome injectable suspension
- Local infiltration with 0.25% bupivacaine with epinephrine (Active Comparator): Patients randomized into the 0.25% bupivacaine with epinephrine group will receive anesthesia and undergo standard posterior spinal fusion surgery under the same condition as the intervention group with one exception: the local infiltration will be made up of equal volume of 0.25% bupivacaine with epinephrine. The equal volume of 0.25% bupivacaine with epinephrine will be used in the exact same administration technique as the liposomal bupivacaine group, involving multiple small-volume injections to the paraspinal musculature spaced approximately 1 centimeter apart.
  Interventions: Drug: Bupivacaine Hydrochloride and Epinephrine Injection

INTERVENTIONS:
Drug: Bupivacaine liposome injectable suspension — EXPAREL is a milky white too off-white aqueous suspension available as single-dose vials. Each mL contains 13.3 mg of bupivacaine, which is contained in multivesicular liposomes.
  Other Names: EXPAREL
  Arms: Local infiltration with liposomal bupivacaine
Drug: Bupivacaine Hydrochloride and Epinephrine Injection — Sensorcaine-MPF with Epinephrine 1:200,000 is a clear, colorless to slightly yellow solution available as single-dose vials. Each mL contains bupivacaine hydrochloride, 0.005 mg epinephrine, and 0.5 mg sodium metabisulfite (antioxidant), and 0.2 mg anhydrous citric acid (stabilizer).
  Other Names: Sensorcaine-MPF with Epinephrine 1:200,000
  Arms: Local infiltration with 0.25% bupivacaine with epinephrine

SUMMARY:
A randomized controlled trial (RCT) investigating whether the local anesthetic injection of liposomal bupivacaine during posterior spinal fusion (PSF) for AIS is more effective in reducing acute postoperative opioid consumption compared to an equal volume injection of 0.25% bupivacaine with epinephrine for patients aged 10 to 17, with 128 patients randomly assigned to one of two arms: liposomal bupivacaine or 0.25% bupivacaine with epinephrine.

ELIGIBILITY:
Inclusion Criteria:

* ≥10 years old and ≤17 years old at assessment
* Diagnosis of Adolescent Idiopathic Scoliosis
* Planned surgical treatment of progressive spinal deformity with posterior spinal fusion

Exclusion Criteria:

* Diagnosis of neuromuscular, syndromic, or congenital scoliosis
* History of known allergy to local anesthesia
* Chronic pre-operative opioid consumptions
* Any other analgesic treatment for chronic pain before surgery
* Psychiatric or neurological disorders
* Cannot fluently read or speak English

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Total amount of morphine equivalents per kilogram | 72 hours postoperatively
  Total amount of morphine equivalents per kilogram during the first 72 hours postoperatively.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) pain scores | 72 hours postoperatively
  The average Numeric Rating Scale pain score (on a scale of 0-10) during the first 72 hours postoperatively will be computed from at most six values typically obtained every four to six hours following surgery. The higher the score, the higher the experienced pain of the individual.
Pain, functional ability, and mental health scores | 1-, 6-, 12-, and 24-months postoperatively
  SRS-22r scores at 1-, 6-, 12-, and 24-months post-operatively. The Scoliosis Patient Questionnaire Version 22r (SRS-22r) is a patient-reported outcome instrument with 22 questions that evaluates the impact of scoliosis and surgery on patient quality of life. Scores from the SRS-22r are compiled into five domain scores: function, pain, self-image, mental health, and satisfaction with management of scoliosis. Each domain score is reported on a scale form 1-5. The lower the score, the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Birch, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No